CLINICAL TRIAL: NCT00290407
Title: Phase II Study of Rituximab Plus B-Glucan in Patients With Chronic Lymphocytic Leukemia(CLL)/Small Lymphocytic Lymphoma (SLL)
Brief Title: Rituximab Plus Beta-Glucan in Chronic Lymphocytic Leukemia(CLL)/Small Lymphocytic Lymphoma (SLL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated due to lack of accrual
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 008.06; BCC-HEM-06-001 (Other: James Graham Brown Cancer Center Clinical Trials Office)
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Leukemia, Lymphocytic, Chronic; Lymphoma, Small Lymphocytic
Keywords: chronic lymphocytic leukemia; small lymphocytic lymphoma; rituximab; beta-glucan
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; beta-Glucans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2, IV (in the vein), once a week for 4 weeks
  Other Names: Rituxan
Dietary Supplement: Beta-Glucan — 250 mg, orally (tablet), three times a day for 9 weeks
  Other Names: Imucell WGP

SUMMARY:
The purpose of this study is to determine how well subjects respond to treatment with Rituximab plus Beta-Glucan.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is the most common form of leukemia in adults. CLL is a cancer of the B-lymphocytes, which make antibodies that help protect the body against harmful foreign substances, such as bacteria and viruses. Similar to CLL, small lymphocytic lymphoma (SLL) is a less-common cancer of the B-lymphocytes. In SLL, the abnormal lymphocytes mainly affect the lymph nodes; in CLL, the abnormal lymphocytes mainly affect the blood and bone marrow.

Current drug therapies for CLL/SLL are known to increase the severity of pre-existing low blood cell counts, which in turn increase the risk of infections in patients. Research to improve the safety and effectiveness of CLL/SLL therapy is currently ongoing. One such therapy being investigated is Rituximab.

Rituximab is a type of drug known as a therapeutic antibody. Therapeutic antibodies are laboratory-created substances that attach onto a protein on the surface of a cell. After binding to the cell, the therapeutic antibody can block the growth of the tumor and/or trigger the body's immune system to attack the target, and can also sensitize a cancer cell to chemotherapy. Rituximab is approved by the Food and Drug Administration (FDA) for the treatment of CLL/SLL.

Beta-Glucan (Imucell WGP) is an over-the-counter dietary supplement that enhances the body's immune system. ImucellTM WGP is extracted from food-grade baker's yeast, which is permitted for use in food by the FDA. Animal studies have shown that Imucell WGP helps trigger the white blood cells to destroy cancer cells. Other animal studies combining Rituximab with Imucell WGP have shown greater tumor regression and tumor-free survival.

ELIGIBILITY:
Inclusion Criteria:

* definitive diagnosis of Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)
* Patients with CLL must have active, progressive, or symptomatic Rai stage II, III, or IV disease. Patients with SLL must have active, progressive or symptomatic stages II, III, IV disease by the Ann Arbor Staging system. Patients with stage I CLL are eligible only if they have systemic symptoms requiring treatment.
* Patients may be treatment naïve, refractory to primary therapy, or relapsed not more than four times) and have measurable or assessable disease. Bone marrow involvement alone will not be acceptable as measurable disease in case of lymphoma.
* Prior therapies may include chemotherapy, radiation, autologous stem cell transplant, or Rituximab.
* Patients who have received therapy must be at least 4 weeks beyond prior standard chemotherapy including corticosteroids, 3 months beyond radiation therapy, and have recovered from significant toxicities from prior therapies
* age > 18 years
* life expectancy of greater than 12 weeks
* ECOG performance status 0, 1, or 2 (Karnofsky > 50%)
* adequate bone marrow function, as defined by: absolute neutrophil count > 1000/µl; platelets > 20,000/µl
* adequate liver function, as defined by: total bilirubin < 2, albumin > 2.5 g/dl, and no ascites; AST(SGOT), ALT(SGPT) & Alkaline Phosphatase < 2.5 x upper limit of normal
* adequate renal function, as defined by: creatinine < 2.5 mg/dl or a creatinine clearance > 30 mL/min (measured or estimated by the Cockcroft-Gault formula) for patients with creatinine levels above 2.5 mg/dl
* must have recovered from acute toxicities resulting from prior therapy to less than grade 1. Alopecia may not be resolved.
* ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study entry or who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* severe autoimmune hemolytic anemia; CNS involvement (either parenchymal or meningeal); severe lymphoma-related symptoms requiring a rapid response to therapy (eg, respiratory compromise due to large effusions or airway obstruction, bowel obstruction, ureteral obstruction, and chylous ascites)
* patients receiving any other investigational agent(s)
* active second malignancy in the last 5 years, except for non-melanoma skin cancer or carcinoma-in-situ
* history of hypersensitivity reactions attributed to Beta-Glucan
* history of connective tissue or autoimmune disease
* patients receiving corticosteroids for any reason, except as a part of treatment for autoimmune hemolytic anemia or immune thrombocytopenia
* uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger H Herzig, MD, Principal Investigator — James Graham Brown Cancer Center/University of Louisville
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

REFERENCES:
- See also: James Graham Brown Cancer Center — http://browncancercenter.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RITUXIMAB PLUS ORAL Β-GLUCAN
Started | 2
Completed | 0
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | RITUXIMAB PLUS ORAL Β-GLUCAN
Number analyzed (Participants) | 2
Age, Customized [Number; unit: participants]
  Over 18 years of age | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: CT Scan to Measure Clinical Effect (Response)
Description: Study terminated, results data not available
Time Frame: 3 months after starting treatment, 6 months after starting treatment, and every 6 months (after completing treatment) until disease progression
Arm/Group | RITUXIMAB PLUS ORAL Β-GLUCAN
Number analyzed (Participants) | 0

2. Secondary Outcome: Blood Specimens Will be Collected to Measure Immunologic Effect
Time Frame: at weeks 4, 8, 12, and at month 6
Arm/Group | RITUXIMAB PLUS ORAL Β-GLUCAN
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | RITUXIMAB PLUS ORAL Β-GLUCAN
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Study terminated, results data not available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No